CLINICAL TRIAL: NCT05800301
Title: Bioretina, Ankara University Technopolis
Brief Title: Management of Retinitis Pigmentosa Via Combination of Wharton's Jelly-derived Mesenchymal Stem Cells and Magnovision
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principal Investigator, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-962-19
Record Dates: First submitted 2023-03-13; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa,; stemcell; Wharton jelly; umbilical cord; mesenchymal stemcell; electromagnetic stimulation; iontophoresis; Magnovision.
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Iontophoresis

STUDY DESIGN:
Intervention Model Description: A total of 130 eyes of 80 RP patients who could be checked regularly, mean 36 months of the follow-up period, were included in this study. Four different groups with similar demographic characteristics were created in the cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Only WJ-MSCs (Active Comparator): Consisted of 34 eyes of 32 RP patients treated with only WJ-MSCs, and it was applied only once following necessary preparations. After the inoculation of stem cells, the patients were followed up regularly on the 10th day, 3rd month, and every 6 months after that until 36 th months. For ethical reasons, the worse eye was selected to inject the stem cells instead of both eyes.
  Interventions: Biological: Wharton's jelly derived mesenchymal stemcells
- Only rEMS (Active Comparator): Consisted of 32 eyes of 16 RP patients treated with only rEMS. rEMS was applied with a custom-designed helmet once a week for 30 min for 36 months. Both eyes are stimulated at the same time with the specially designed system for ophthalmologic use (MagnoVisionTM).
  Interventions: Device: Magnovision
- WJ-MSCs and rEMS combination (Active Comparator): Consisted of 32 eyes of 16 RP patients treated with the WJ-MSCs and rEMS combination. WJ-MSCs were applied first into the deep subtenon space of both eyes after necessary preparations. rEMS application was started 10 days after the WJ-MSC application with a custom-designed helmet for 30 min. WJ-MSCs were inoculated only once, and rEMS was applied regularly once a week for 30 min for 36 months. Both eyes are stimulated at the same time with the specially designed system for ophthalmologic use (MagnoVisionTM).
  Interventions: Biological: Wharton's jelly derived mesenchymal stemcells; Device: Magnovision
- The natural course (No Intervention): The natural course (control) group consisted of 32 eyes of 16 RP patients who received no treatment and were regularly followed until the 36th month. This group comprised patients who did not accept any treatment and/or were in good condition at baseline.

INTERVENTIONS:
Biological: Wharton's jelly derived mesenchymal stemcells — The WJ-MSCs suspension from the culture was delivered to the operating room by cold chain and used within 24 h. A total of 1.5 ml of the WJ-MSC suspension was immediately injected into the deep subtenon space of each eye.
  Arms: Only WJ-MSCs; WJ-MSCs and rEMS combination
Device: Magnovision — Specifically designed helmets producing high-frequency repetitive electromagnetic stimulation (MagnovisionTM, Bioretina Biotechnology, Ankara, Türkiye) stimulated the retinas and visual pathways in both eyes.
  Other Names: Electromagnetic stimulator; iontophoresis; neuromodulator
  Arms: Only rEMS; WJ-MSCs and rEMS combination

SUMMARY:
Purpose To investigate whether the natural progression rate of retinitis pigmentosa (RP) can be decreased with subtenon umbilical cord Wharton's jelly derived mesenchymal stemcell (WJ-MSC) application alone or combination with retinal electromagnetic stimulation (rEMS).

Material and methods The study included prospective analysis of 130 eyes of 80 retinitis pigmentosa patients with a 36-month follow-up duration. Patients constitute 4 groups with similar demographic characteristics. The subtenon WJ-MSC only group consisted of 34 eyes of 32 RP patients as Group1; The rEMS only group consisted of 32 eyes of 16 RP patients as Group2; The combined management group consisted of 32 eyes of 16 RP patients who received combined WJ-MSC and rEMS as Group3; The natural course (control) group consisted of 32 eyes of 16 RP patients who did not receive any treatment were classified as Group4. Fundus autofluorescence surface area (FAF-field), horizontal and vertical ellipsoid zone width (EZW), fundus perimetry deviation index (FPDI), full field electroretinography magnitude (ERG-m) and best corrected visual acuity (BCVA) changes were compared within and between groups after 36 month follow up period.

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP) is one of the most common inherited diseases of retinopathies. It is estimated to affect 1 in 3000 to 1 in 4000 people globally. Retinitis pigmentosa (RP) is a genetic disease group characterized by progressive loss of photoreceptors. At least 90 different structural and functional proteins have been identified in the sensory retina, which is necessary for the healthy functioning of the visual cycle. At least 300 genes encode these proteins, and their fragments have been identified in the sensory retina. Mutations in any of these 300 genes lead to outer retinal degeneration and RP. In classical RP, genetic mutations primarily impair the functions of rod cells. Structural and functional protein deficiency causes rod cells to enter the dormant phase and undergo apoptosis. The inheritance pattern can be autosomal dominant, autosomal recessive, X-linked, mitochondrial, or spontaneous mutations. The rate of disease progression is different in each inheritance pattern. Patients first complain of difficulty seeing at night and prolonged dark adaptation. As rod cell loss increases, the peripheral visual field begins to narrow. The narrowing of the visual field progresses at a rate of 5-15% each year, depending on the inheritance pattern, and finally, the cone cells are affected. Apoptosis of rod/cone cells results in end-stage RP, then progress to total blindness.

Wharton's jelly-derived mesenchymal stem cells (WJ-MSCs) have a high paracrine effect and secrete exosomes containing different growth factors (GFs) and neurotrophins. These peptides in the exosome content are functional and structural peptides for neurons. Peptides that cannot be encoded in RP can be substituted by WJ-MSCs exosomes. Growth factors and neurotrophins in the exosome can accelerate the entry of glucose into retina pigment epithelium (RPE) and photoreceptors and their conversion to ATP, an energy molecule. These neurotrophins can also provide homeostasis, preventing apoptosis by accelerating the phagocytosis of cellular metabolic wastes.

High-frequency repetitive electromagnetic stimulation (rEMS) can modulate ion channels in neurons depending on frequency, magnetic field, and duration variables. If the dormant phase - which is the sleep mode caused by genetic mutations in the sensory retina - is prolonged, apoptosis and permanent photoreceptor loss occur. Activation of ion channels and acceleration of neuromodulation by electromagnetic stimulation can prevent neuronal apoptosis. Scientific studies have also shown that rEMS increases mesenchymal stem cells' exosome degranulation. Another effect of rEMS is the iontophoresis effect. The passage of large molecules into the cells through the scleral pores is possible by changing the electrical charges between neurotrophins and their receptors and increasing the affinity. It can also induce the delivery of higher amounts of GFs and neurotrophins into the subretinal environment and retina.

This prospective clinical study aims to investigate whether RP progression can be slowed or maintained with the inoculation of WJ-MSCs alone into the deep subtenon space or in conjunction with rEMS application compared to the natural course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* RP patients of any genotype and phenotype;
* BCVA better than 35 letters;
* Any degree and kind of visual field loss;
* Over 18 years old.

Exclusion Criteria:

* The presence of glaucoma,
* Dense cataracts
* Dense vitreus opacities
* Autoimmune retinopathy-like clinical picture
* Any degree of smoking
* Presence of systemic neurological disease with seizure
* Presence of a cardiac pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fundus autofluorescence surface area (FAF-field): | Change between the 36th month (Time1) and baseline (Time0) values.
  The pattern of FAF correlates well with functional tests such as perimetry and ERG. The ring of increased autofluorescence appears to represent the border between functional and dysfunctional retinas. Metabolically active photoreceptors/RPE appear as hyperfluorescent areas in the FAF device due to the presence of lipofuscin. The FAF device calculated the FAF field automatically after marking the horizontal and vertical longest axes of the hyperfluorescent field in the posterior pole.

SECONDARY OUTCOMES:
ETDRS visual acuity (BCVA): | Change between the 36th month (Time1) and baseline (Time0) values.
  The visual acuity scores obtained from the T0 and T1 examinations were analyzed and compared using statistical tests to determine effectiveness.
Ellipsoid zone widths (EZW): | Change between the 36th month (Time1) and baseline (Time0) values.
  EZW showed healthy photoreceptors and was measured horizontally and vertically (HEZW and VEZW, respectively) on multimodal OCTA devices. A manual segmentation program was used for the measurement of EZW.
Fundus perimetry deviation index (FPDI): | Change between the 36th month (Time1) and baseline (Time0) values.
  FPDI records were examined in the 24/2 visual field (VF) of the computerized perimetry records. The FPDI offers data explaining how many of the 100 flashing points and what percentage of the visual field could be correctly seen by the patient. For VF analysis, practice rounds were carried out three times before the last assessments to avoid mistakes during the test.
Full-ﬁeld multi-luminance flicker electroretinography magnitude (ERG-m): | Change between the 36th month (Time1) and baseline (Time0) values.
  Digital electroretinography is a non-invasive office-based objective test that measures the electrical activity of the global outer retinal cells in response to a light stimulus. ERG-m refers to the action potentials and phase deviations recorded from photoreceptors stimulated with different light intensities.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - BioRetina, Ankara, Gölbaşı
  - Ankara University Biotechnology Institute, Ankara, Türkiye
  - Umut Arslan, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozmert E, Arslan U. Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet-Rich Plasma: Preliminary Clinical Results. Adv Ther. 2019 Sep;36(9):2273-2286. doi: 10.1007/s12325-019-01040-2. Epub 2019 Aug 5. PMID 31385285
- [Background] Arslan U, Ozmert E. Treatment of resistant chronic central serous chorioretinopathy via platelet-rich plasma with electromagnetic stimulation. Regen Med. 2020 Aug;15(8):2001-2014. doi: 10.2217/rme-2020-0056. Epub 2020 Oct 27. PMID 33107400
- [Result] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872
- [Result] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly-derived mesenchymal stem cells: prospective analysis of 1-year results. Stem Cell Res Ther. 2020 Aug 12;11(1):353. doi: 10.1186/s13287-020-01870-w. PMID 32787913
- [Result] Ozmert E, Arslan U. Management of toxic optic neuropathy via a combination of Wharton's jelly-derived mesenchymal stem cells with electromagnetic stimulation. Stem Cell Res Ther. 2021 Sep 27;12(1):518. doi: 10.1186/s13287-021-02577-2. PMID 34579767
- [Result] Arslan U, Ozmert E. Management of Retinitis Pigmentosa via Platelet-Rich Plasma or Combination with Electromagnetic Stimulation: Retrospective Analysis of 1-Year Results. Adv Ther. 2020 May;37(5):2390-2412. doi: 10.1007/s12325-020-01308-y. Epub 2020 Apr 18. PMID 32303913
- [Derived] Ozmert E, Arslan U. Management of Retinitis Pigmentosa Via Wharton's Jelly-Derived Mesenchymal Stem Cells or Combination With Magnovision: 3-Year Prospective Results. Stem Cells Transl Med. 2023 Oct 5;12(10):631-650. doi: 10.1093/stcltm/szad051. PMID 37713598